CLINICAL TRIAL: NCT00523861
Title: The Effect of Moderate Alcohol Consumption on Glucose Metabolism and Gastric Emptying in Healthy, Lean and Overweight Young Men
Brief Title: Moderate Alcohol Consumption, Glucose Metabolism and Gastric Emptying
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TNO (Other)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: P6281; Alcohol Research 19
Record Dates: First submitted 2007-08-30; First posted 2007-09-03 (Estimated); Last update posted 2007-09-14 (Estimated); Status verified 2007-08

CONDITIONS: Lean; Obese
Keywords: Glucose; Insulin sensitivity; Glucose metabolism; Appetite; Satiety
MeSH Terms: conditions — Obesity; Insulin Resistance | interventions — Ethanol; Economics

INTERVENTIONS:
Dietary Supplement: Moderate alcohol consumption

SUMMARY:
Moderate alcohol consumption is associated with a decreased risk of type II diabetes mellitus. In a recent study of Greenfield et al. it was observed that moderate alcohol consumption significantly improved postprandial glucose concentrations. Similar observations were made in our previous study. One of the mechanisms by which this may occur is delayed gastric emptying after alcohol consumption.

DETAILED DESCRIPTION:
Purpose: The primary objective of this study is to investigate the effect of moderate daily alcohol consumption on hepatic glucose uptake and peripheral glucose storage. Secondly, the effect of moderate alcohol consumption on gastric emptying and postprandial wellness will be studied. These effects will be studied in apparently healthy, lean or overweight young men.

Design: Randomized, partially diet-controlled, placebo controlled cross-over design.

Subjects: Healthy male lean and obese volunteers aged between 18 and 40 years (n=18).

Intervention: During 2 periods of 21 days either white wine or white grape juice has to be consumed with the evening meal. The last 7 days of each period will be fully dietary controlled.

Treatment A: 375 ml of white wine (35 g alcohol) per day Treatment B: 375 ml of white grape juice per day

Measures:

* Glucose metabolism: glucose uptake and peripheral glucose storage (measurement of isotopic enriched plasma glucose levels.
* Gastric emptying and postprandial wellness.
* Postprandial glycemic response and related factors (glucose, insulin, lactate, FFA, glucagon, ghrelin, CCK, GIP, GLP-1, PYY, triglycerides, total cholesterol, HDL cholesterol, LDL cholesterol, paracetamol (absorption test)

ELIGIBILITY:
Inclusion Criteria:

* Healthy as assessed by the:
* physical examination
* results of the pre-study laboratory tests
* Males aged between 18 and 40 years at Day 01 of the study (including 18 and 40)
* Lean subjects and overweight/obese subjects: BMI 18.5-35 kg/m2
* Alcohol consumption between 7 and 28 units/week (including 7 and 28)
* Non restrained eater, defined as a score ≤ 2.5 on the Dutch Restrained Eating Questionnaire

Exclusion Criteria:

* Smoking
* Not willing or able to change habitual alcohol consumption during the study according to protocol
* Having an allergy for paracetamol

Ages: 18 Years to 40 Years | Sex: Male
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2005-05; Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to investigate the effect of moderate daily alcohol consumption on hepatic glucose uptake and peripheral glucose storage | 3 weeks

SECONDARY OUTCOMES:
Secondly, the effect of moderate alcohol consumption on gastric emptying and postprandial wellness will be studied. | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Henk FJ Hendriks, PhD, Principal Investigator — Hendriks HFJ
Locations (1):
- TNO Quality of Life, Zeist, Utrecht, Netherlands